CLINICAL TRIAL: NCT00150618
Title: A Phase III, Randomized, Double-Blind, Multi-Center, Parallel-Group, Placebo-Controlled Safety and Efficacy Study of SPD503 in Children and Adolescents Aged 6-17 With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Safety and Efficacy of SPD503 in Treating ADHD in Children and Adolescents Aged 6-17
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPD503-304
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2009-10-15 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Guanfacine

ARMS (5):
- SPD503 (Guanfacine HCl) (1 mg) (Experimental)
  Interventions: Drug: SPD503 (1 mg)
- SPD503 (2 mg) (Experimental)
  Interventions: Drug: SPD503 (2 mg)
- SPD503 (3 mg) (Experimental)
  Interventions: Drug: SPD503 (3 mg)
- SPD503 (4 mg) (Experimental)
  Interventions: Drug: SPD503 (4 mg)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPD503 (1 mg)
  Other Names: Guanfacine hydrochloride
  Arms: SPD503 (Guanfacine HCl) (1 mg)
Drug: SPD503 (2 mg)
  Arms: SPD503 (2 mg)
Drug: SPD503 (3 mg)
  Arms: SPD503 (3 mg)
Drug: SPD503 (4 mg)
  Arms: SPD503 (4 mg)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of SPD503 compared to placebo in the treatment of children and adolescents aged 6-17 with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a primary diagnosis of ADHD
* Females of childbearing potential must have a negative serum beta human chorionic gonadotropin (HCG) pregnancy test
* Male or non-pregnant female subject who agrees to comply with any applicable contraceptive requirements

Exclusion Criteria:

* Subject has a current, uncontrolled, comorbid psychiatric diagnosis with significant symptoms such as severe comorbid Axis II disorders or severe Axis I disorders
* Subject weighs less than 55 lbs or is morbidly overweight with a BMI => 35
* Subject has a history of seizure during the last 2 years or a serious tic disorder, including Tourette's Disorder
* Subject is pregnant or lactating

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 324 (Actual)
Dates: Start 2004-03-30 (Actual); Primary Completion 2004-10-07 (Actual); Study Completion 2004-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

REFERENCES:
- [Result] Sallee FR, McGough J, Wigal T, Donahue J, Lyne A, Biederman J; SPD503 STUDY GROUP. Guanfacine extended release in children and adolescents with attention-deficit/hyperactivity disorder: a placebo-controlled trial. J Am Acad Child Adolesc Psychiatry. 2009 Feb;48(2):155-65. doi: 10.1097/CHI.0b013e318191769e. PMID 19106767
- See also: FDA recall information — http://www.fda.gov/opacom/7alerts.html
- See also: FDA-approved label — http://www.intuniv.com/documents/INTUNIV_Full_Prescribing_Information.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although 324 subjects were randomized, 2 never received drug and therefore were not included in the Baseline Characteristics. Subjects received either 1, 2, 3, or 4 mg of SPD503 (Guanfacine hydrochloride) or placebo once daily.
Groups:
- SPD503 (1 mg); SPD503 (2 mg); SPD503 (3 mg); SPD503 (4 mg): Guanfacine HCl once daily
- Placebo: once daily
Period: Overall Study
Arm/Group | SPD503 (1 mg) | SPD503 (2 mg) | SPD503 (3 mg) | SPD503 (4 mg) | Placebo
Started | 62 | 65 | 65 | 66 | 66
Completed | 45 | 47 | 38 | 40 | 41
Not Completed | 17 | 18 | 27 | 26 | 25
Not completed — Adverse Event | 2 | 2 | 6 | 9 | 5
Not completed — Withdrawal by Subject | 6 | 8 | 8 | 4 | 5
Not completed — Lost to Follow-up | 4 | 1 | 5 | 8 | 4
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 1 | 4 | 7 | 4 | 6
Not completed — No study meds | 0 | 0 | 0 | 0 | 2
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 1
Not completed — Lack of compliance | 2 | 1 | 1 | 0 | 1
Not completed — Abnormal ECG | 1 | 0 | 0 | 0 | 0
Not completed — Sponsor's decision | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SPD503 (1 mg) | SPD503 (2 mg) | SPD503 (3 mg) | SPD503 (4 mg) | Placebo | Total
Number analyzed (Participants) | 61 | 65 | 65 | 65 | 66 | 322
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 61 | 65 | 65 | 65 | 66 | 322
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.3 (2.14) | 10.6 (2.81) | 11.1 (2.96) | 10.5 (2.53) | 10.8 (2.89) | 10.5 (2.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 19 | 17 | 12 | 21 | 89
  Male | 41 | 46 | 48 | 53 | 45 | 233
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 61 | 65 | 65 | 65 | 66 | 322

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-RS-IV) Score at 6 Weeks
Description: Change in the Attention Deficit Hyperactivity Disorder Rating Scale-fourth edition (ADHD-RS-IV) total score from baseline. The ADHD-RS-IV consists of 18 items scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with total score ranging from 0 to 54.
Time Frame: Baseline and 6 weeks
Population: Intent to treat (ITT) defined as all subjects who were randomized to treatment and had the Baseline and at least one post-randomization primary efficacy measurement.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | SPD503 (1 mg) | SPD503 (2 mg) | SPD503 (3 mg) | SPD503 (4 mg) | Placebo
Number analyzed (Participants) | 57 | 63 | 60 | 63 | 63
Units on a Scale | -19.44 (1.69) | -18.09 (1.60) | -20.00 (1.64) | -20.57 (1.60) | -12.69 (1.60)
Statistical Analysis 1: Comparison: SPD503 (1 mg) vs Placebo; Test type: Superiority or Other; p = 0.0041, ANCOVA
Statistical Analysis 2: Comparison: SPD503 (2 mg) vs Placebo; Test type: Superiority or Other; p = 0.0176, ANCOVA
Statistical Analysis 3: Comparison: SPD503 (3 mg) vs Placebo; Test type: Superiority or Other; p = 0.0016, ANCOVA
Statistical Analysis 4: Comparison: SPD503 (4 mg) vs Placebo; Test type: Superiority or Other; p = 0.0006, ANCOVA

2. Secondary Outcome: Change From Baseline in Conner's Parent Rating Scale-revised Short Version (CPRS-R) Score at 6 Weeks
Description: The Conner's Parent rating Scale-revised short version (CPRS-R) consists of 27 questions graded on a scale from 0 (not true at all) to 3 (very much true) with a total score ranging from 0 to 81. Higher scores are indicative of increased ADHD. This scale allows parents to respond on the basis of the child's behavior and help assess ADHD and evaluate problem behavior.
Time Frame: Baseline and 6 weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | SPD503 (1 mg) | SPD503 (2 mg) | SPD503 (3 mg) | SPD503 (4 mg) | Placebo
Number analyzed (Participants) | 52 | 55 | 47 | 53 | 53
Units on a Scale | -19.50 (2.36) | -14.96 (2.29) | -17.94 (2.48) | -15.93 (2.34) | -8.41 (2.34)
Statistical Analysis 1: Comparison: SPD503 (1 mg) vs Placebo; Test type: Superiority or Other; p = 0.0010, ANCOVA
Statistical Analysis 2: Comparison: SPD503 (2 mg) vs Placebo; Test type: Superiority or Other; p = 0.0468, ANCOVA
Statistical Analysis 3: Comparison: SPD503 (3 mg) vs Placebo; Test type: Superiority or Other; p = 0.0056, ANCOVA
Statistical Analysis 4: Comparison: SPD503 (4 mg) vs Placebo; Test type: Superiority or Other; p = 0.0237, ANCOVA

3. Secondary Outcome: Number of Participants With Improvement in Clinical Global Impression-Improvement (CGI-I)
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: 6 weeks
Population: ITT
Measure: Number; unit: Participants
Arm/Group | SPD503 (1 mg) | SPD503 (2 mg) | SPD503 (3 mg) | SPD503 (4 mg) | Placebo
Number analyzed (Participants) | 57 | 63 | 60 | 63 | 63
Participants | 31 | 27 | 33 | 35 | 19
Statistical Analysis 1: Comparison: SPD503 (1 mg) vs Placebo; Test type: Superiority or Other; p = 0.0074, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: SPD503 (2 mg) vs Placebo; Test type: Superiority or Other; p = 0.1404, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: SPD503 (3 mg) vs Placebo; Test type: Superiority or Other; p = 0.0055, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: SPD503 (4 mg) vs Placebo; Test type: Superiority or Other; p = 0.0041, Cochran-Mantel-Haenszel

4. Secondary Outcome: Number of Participants With Improvement in Parent Global Assessment (PGA)
Description: Parent Global Assessment (PGA) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: 6 weeks
Population: ITT
Measure: Number; unit: Participants
Arm/Group | SPD503 (1 mg) | SPD503 (2 mg) | SPD503 (3 mg) | SPD503 (4 mg) | Placebo
Number analyzed (Participants) | 53 | 55 | 47 | 53 | 53
Participants | 27 | 20 | 29 | 30 | 16
Statistical Analysis 1: Comparison: SPD503 (1 mg) vs Placebo; Test type: Superiority or Other; p = 0.0303, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: SPD503 (2 mg) vs Placebo; Test type: Superiority or Other; p = 0.4982, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: SPD503 (3 mg) vs Placebo; Test type: Superiority or Other; p = 0.0017, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: SPD503 (4 mg) vs Placebo; Test type: Superiority or Other; p = 0.0063, Cochran-Mantel-Haenszel

5. Secondary Outcome: Change From Baseline in Child Health Questionnaire-Parent Form (CHQ-PF50) Score at 6 Weeks
Description: The Child Health Questionnaire-Parent Form (CHQ-PF50) was developed to measure the physical and psychosocial well-being of children aged 5 years of age and older. Total scoring ranges from 0-100. Increases in scores represent improved well-being in subjects as assessed by their parents.
Time Frame: Baseline and 6 weeks
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | SPD503 (1 mg) | SPD503 (2 mg) | SPD503 (3 mg) | SPD503 (4 mg) | Placebo
Number analyzed (Participants) | 48 | 45 | 37 | 40 | 42
units on a scale
  Physical | 0.32 (0.87) | 0.35 (0.89) | -0.91 (0.99) | -2.44 (0.95) | -0.01 (0.92)
  Psychosocial | 10.61 (1.41) | 7.47 (1.44) | 9.07 (1.61) | 9.43 (1.53) | 6.34 (1.49)
Statistical Analysis 1: Comparison: SPD503 (1 mg) vs Placebo; Psychosocial category; Test type: Superiority or Other; p = 0.0383, ANCOVA
Statistical Analysis 2: Comparison: SPD503 (2 mg) vs Placebo; Psychosocial category; Test type: Superiority or Other; p = 0.5859, ANCOVA
Statistical Analysis 3: Comparison: SPD503 (3 mg) vs Placebo; Psychosocial category; Test type: Superiority or Other; p = 0.2136, ANCOVA
Statistical Analysis 4: Comparison: SPD503 (4 mg) vs Placebo; Psychosocial category; Test type: Superiority or Other; p = 0.1483, ANCOVA

ADVERSE EVENTS:
Arm/Group | SPD503 (1 mg) | SPD503 (2 mg) | SPD503 (3 mg) | SPD503 (4 mg) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/65 | 1/65 | 0/65 | 1/66
Other Adverse Events (participants affected / at risk) | 49/61 | 40/65 | 45/65 | 55/65 | 45/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPD503 (1 mg) (N=61) | SPD503 (2 mg) (N=65) | SPD503 (3 mg) (N=65) | SPD503 (4 mg) (N=65) | Placebo (N=66)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SPD503 (1 mg) (N=61) | SPD503 (2 mg) (N=65) | SPD503 (3 mg) (N=65) | SPD503 (4 mg) (N=65) | Placebo (N=66)
Upper abdominal pain (Gastrointestinal disorders) | 5 | 2 | 1 | 8 | 6
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 5 | 1
Nausea (Gastrointestinal disorders) | 4 | 2 | 3 | 4 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 3 | 1 | 4
Fatigue (General disorders) | 6 | 3 | 7 | 8 | 2
Lethargy (General disorders) | 1 | 0 | 5 | 3 | 1
Dizziness (Nervous system disorders) | 3 | 0 | 6 | 6 | 4
Headache (Nervous system disorders) | 16 | 16 | 5 | 16 | 7
Sedation (Nervous system disorders) | 1 | 6 | 3 | 5 | 3
Somnolence (Nervous system disorders) | 16 | 11 | 15 | 27 | 8
Irritability (Psychiatric disorders) | 4 | 4 | 2 | 4 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2 | 1 | 0
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 1 | 4
Hypotension (Vascular disorders) | 2 | 1 | 4 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.